CLINICAL TRIAL: NCT03762824
Title: Combined Pneumococcal Conjugate and Polysaccharide Vaccination in Inflammatory Rheumatic Disease. Impact of Antirheumatic Treatment on Antibody Response.
Brief Title: Combined Pneumococcal Conjugate and Polysaccharide Vaccination in Inflammatory Rheumatic Disease
Acronym: IPS-BOOSTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPS-BOOSTER
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus; Sjögren Syndrome; Systemic Vasculitis; Spondyloarthritis
Keywords: Pneumococcal Conjugate Vaccine; Pneumococcal Disease; Immune Response; Inflammatory Rheumatic Disease; Pneumococcal Polysaccharide Vaccine; Immunosuppression
MeSH Terms: conditions — Arthritis, Rheumatoid; Sjogren's Syndrome; Systemic Vasculitis; Spondylarthritis; Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- PCV13+PPV23 vaccinated patients (Active Comparator): Patients with different inflammatory rheumatic diseases are immunized with one dose 13-valent pneumococcal conjugate vaccine 0.5 ml i.m., followed by one dose 23-valent pneumococcal polysaccharide vaccine 0.5 ml i.m. after 8 weeks.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: 23-valent pneumococcal polysaccharide vaccine
- PCV13+PPV23 vaccinated controls (Active Comparator): Healthy controls are immunized with one dose 13-valent pneumococcal conjugate vaccine 0.5 ml i.m., followed by one dose 23-valent pneumococcal polysaccharide vaccine 0.5 ml i.m. after 8 weeks.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: 23-valent pneumococcal polysaccharide vaccine
- PPV23-booster to previous PCV-vaccinated patients (Active Comparator): Patients with different inflammatory rheumatic disease previously immunized with one dose PCV7 or PCV13 within another study (see VACCIMIL), are immunized with one dose PPV23 0.5 ml i.m.
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- PCV13 to previous PPV23-vaccinated patients (Active Comparator): Patients with different inflammatory rheumatic disease previously immunized with one dose PPV23 within another study (see VACCIMIL), are immunized with one dose PCV13 0.5 ml i.m.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- PPV23-booster to previous PCV-vaccinated controls (Active Comparator): Healthy controls previously immunized with one dose PCV7 or PCV13 within another study (see VACCIMIL), are immunized with one dose PPV23 0.5 ml i.m.
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Pneumococcal conjugate vaccination during antirheumatic treatment
  Other Names: Prevenar 13; PCV13
  Arms: PCV13 to previous PPV23-vaccinated patients; PCV13+PPV23 vaccinated controls; PCV13+PPV23 vaccinated patients
Biological: 23-valent pneumococcal polysaccharide vaccine — Pneumococcal polysaccharide vaccination during antirheumatic treatment
  Other Names: Pneumovax; PPV23
  Arms: PCV13+PPV23 vaccinated controls; PCV13+PPV23 vaccinated patients; PPV23-booster to previous PCV-vaccinated controls; PPV23-booster to previous PCV-vaccinated patients

SUMMARY:
The overall objective of this project is to study the influence of modern anti-inflammatory treatments in established inflammatory rheumatic diseases (IRD) on antibody response elicited by pneumococcal vaccination using 13-valent conjugate vaccine in combined schedules with 23-valent polysaccharide vaccine. In addition, the aim is to study the clinical aspects of vaccination regarding: tolerability in immunosuppressed patients with IRD, impact on existing rheumatic disease, possible association with onset of new autoimmune diseases, long-term immunity following pneumococcal vaccination and efficacy in preventing invasive pneumococcal disease. Results from this study are expected to bridge the existing knowledge gap and contribute to body of evidence needed for recommendations and implementation of vaccination program in IRD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with IRD receiving active anti-rheumatic treatments with DMARDs or biological remedies are offered to participate in the study. The protocol permits stratification for prednisolone usage.

Exclusion Criteria:

* known allergy/intolerance of pneumococcal vaccine
* pregnancy
* active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
2-fold rise in pneumococcal serotype-specific antibody concentration | 8 weeks after pneumococcal conjugate vaccine and 4-6 weeks after polysaccharide vaccination
  Pneumococcal serotype-specific antibody concentration (12-valent)

SECONDARY OUTCOMES:
Functional antibody response | 8 weeks after pneumococcal conjugate vaccine and 4-6 weeks after polysaccharide vaccination
  Opsonophagocytosis activity assay
Long-term serotype-specific immunity to pneumococcal disease | 3 years after vaccination
  Pneumococcal serotype-specific antibody concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jehns Martineus, MD, Study Director — Skåne Universitets sjukhus, dept of rheumatology

IPD SHARING:
Plan to Share IPD: Undecided
If requested we will consider sharing unidentified individual patient data

REFERENCES:
- [Background] Doran MF, Crowson CS, Pond GR, O'Fallon WM, Gabriel SE. Frequency of infection in patients with rheumatoid arthritis compared with controls: a population-based study. Arthritis Rheum. 2002 Sep;46(9):2287-93. doi: 10.1002/art.10524. PMID 12355475
- [Background] Kapetanovic MC, Saxne T, Sjoholm A, Truedsson L, Jonsson G, Geborek P. Influence of methotrexate, TNF blockers and prednisolone on antibody responses to pneumococcal polysaccharide vaccine in patients with rheumatoid arthritis. Rheumatology (Oxford). 2006 Jan;45(1):106-11. doi: 10.1093/rheumatology/kei193. Epub 2005 Nov 15. PMID 16287919
- [Background] Kapetanovic MC, Roseman C, Jonsson G, Truedsson L, Saxne T, Geborek P. Antibody response is reduced following vaccination with 7-valent conjugate pneumococcal vaccine in adult methotrexate-treated patients with established arthritis, but not those treated with tumor necrosis factor inhibitors. Arthritis Rheum. 2011 Dec;63(12):3723-32. doi: 10.1002/art.30580. PMID 21834061
- [Background] Nived P, Nagel J, Saxne T, Geborek P, Jonsson G, Skattum L, Kapetanovic MC. Immune response to pneumococcal conjugate vaccine in patients with systemic vasculitis receiving standard of care therapy. Vaccine. 2017 Jun 22;35(29):3639-3646. doi: 10.1016/j.vaccine.2017.05.044. Epub 2017 May 25. PMID 28552512
- [Background] Centers for Disease Control and Prevention (CDC). Use of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal polysaccharide vaccine for adults with immunocompromising conditions: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Morb Mortal Wkly Rep. 2012 Oct 12;61(40):816-9. PMID 23051612
- [Derived] Nived P, Jonsson G, Settergren B, Einarsson J, Olofsson T, Jorgensen CS, Skattum L, Kapetanovic MC. Prime-boost vaccination strategy enhances immunogenicity compared to single pneumococcal conjugate vaccination in patients receiving conventional DMARDs, to some extent in abatacept but not in rituximab-treated patients. Arthritis Res Ther. 2020 Feb 22;22(1):36. doi: 10.1186/s13075-020-2124-3. PMID 32087733